CLINICAL TRIAL: NCT00072787
Title: A Phase I/II, Open-Label, Nonrandomized, Dose-Finding Safety, Tolerance, Pharmacokinetic, and Efficacy Study of Orally Administered S-1 in Combination With Cisplatin in Patients With Advanced Gastric Cancer
Brief Title: Phase 1/2 Study of S-1 and Cisplatin in Advanced Gastric Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Taiho Oncology, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPU-S1101; ID02-694
Record Dates: First submitted 2003-11-10; First posted 2003-11-13 (Estimated); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; phase 2 clinical trial
MeSH Terms: conditions — Stomach Neoplasms | interventions — S 1 (combination); Cisplatin

INTERVENTIONS:
Drug: S-1
Drug: cisplatin

SUMMARY:
The purpose of the phase 1 portion of the study is to determine the safe dose of S-1 and cisplatin that can be administered in gastric cancer patients.

The purpose of the phase 2 portion of the study is to determine the antitumor activity of the S-1 and cisplatin regimen established from phase 1 in patients with advanced gastric cancer.

DETAILED DESCRIPTION:
S-1 is an oral fluoropyrimidine which combines tegafur (a 5-FU prodrug) with two classes of modulators which:

* inhibit dihydropyrimidine dehydrogenase (DPD) and
* block phosphorylation of 5-FU in gastrointestinal tissues.

S-1 is designed to enhance the the clinical utility of an oral fluoropyrimidine while ameliorating the disadvantage of gastrointestinal toxicity.

5-Fu and cisplatin have been used as a standard treatment in gastric cancer and preliminary data indicate that S-1 plus cisplatin may result in superior tolerability and efficacy in advanced gastric cancer.

S-1 is currently approved in Japan for treatment of gastric cancer and head and neck cancer.

ELIGIBILITY:
Inclusion Criteria

* Has histologically or cytologically confirmed adenocarcinoma of the stomach or gastroesophageal junction
* Has advanced, unresectable cancer at the time of study entry
* Has measurable disease as defined by RECIST criteria, i.e., lesions that can be accurately measured in at least one dimension with the longest diameter ≥20 mm using conventional techniques or ≥10 mm using spiral CT scan
* Is at least 3 weeks post-gastrectomy surgery
* Has not received prior chemotherapy for their cancer (adjuvant therapy is permitted and does not count as prior chemotherapy).
* Has performance status of ≥ 70% on the Karnofsky scale (Appendix B)
* Has a predicted life expectancy of ≥ 12 weeks
* Has an absolute granulocyte count of ≥ 1,500/mm3
* Has a platelet count ≥ 100,000/mm3
* Has a hemoglobin of ≥ 9.0 g/dL
* Has a bilirubin of ≤ 1.5 times the ULN
* Has transaminases ≤ 2.5 times the ULN except for patients with liver metastasis who may have transaminases ≤ 5 times the ULN
* Has a creatinine ≤ ULN and calculated creatinine ≥ 60 mL/min
* According to the judgment of the Investigator, the patient has recovered from all previous anti-cancer treatment-related toxicities to at least Grade 1 (see exceptions above)
* Has stopped all previous investigational drugs at least 4 weeks prior to treatment with S-1 and cisplatin.
* Is able to take medications orally
* Female patients of childbearing potential who are not pregnant and who use acceptable means of contraception while on study and for an additional 30 days after the last dose of study medication. Male patients must use adequate contraception.

Exclusion Criteria

* Has relapsed within 6 months from the end of adjuvant therapy
* Has known brain or leptomeningeal metastases.
* Has any other serious illness or medical condition(s) including, but not limited to, the following:

  * uncontrolled congestive heart failure, angina pectoris, arrhythmias, or hypertension ; or any significant medical condition that is a contraindication for chemotherapy
  * concurrent malignancy other than gastric cancer except adequately treated carcinoma-in-situ of the cervix or non-melanoma skin cancer
  * active infection
  * gastrointestinal disorder, including malabsorption, chronic nausea and vomiting, chronic diarrhea
  * unstable diabetes mellitus
  * psychiatric disorder that may interfere with consent and/or protocol compliance
  * known neuropathy (including hearing loss) at baseline of Grade 2 or higher (as per NCI CTC v2.0 see Appendix A)
* Has known hypersensitivity to any of the constituents of the study medication
* Is receiving a concomitant treatment with drugs interacting with S-1.
* Is a pregnant or lactating female or who refuses to use an acceptable means of contraception. Is a male and refuses to use an acceptable means of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41
Dates: Start 2003-10; Primary Completion 2006-03 (Actual); Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Rosen, Lee, Los Angeles, California
  - University of Southern California Norris Comprehensive Cancer Center, Los Angeles, California
  - Chong, Clayton, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - Northwestern University Robert H Lurie Comprehensive Cancer Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Lovelace Sandia Health System, Albuquerque, New Mexico
  - New Mexico VA Health Care System, Albuquerque, New Mexico
  - University of New Mexico - Albuquerque, Albuquerque, New Mexico
  - Abramson Cancer Center at the University of Pennsylvania, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas